CLINICAL TRIAL: NCT01902446
Title: A Pilot Study of Prehospital Oral Chlorhexidine Gluconate to Prevent Early Ventilator Associated Pneumonia in Intubated Trauma Patients
Brief Title: Prehospital Ventilator-Associated Pneumonia Prevention Trial
Acronym: P-VAPP
Status: Completed | Type: Observational
Sponsor: Nicholas M Mohr (Other)
Responsible Party: Sponsor-Investigator, Nicholas M Mohr, Assistant Professor of Emergency Medicine and Anesthesia Critical Care, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201304766
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Wounds and Injuries; Respiratory Failure; Pneumonia, Ventilator-Associated
Keywords: Chlorhexidine; Randomized Controlled Trial; Emergency Medical Services; Intubation, Endotracheal
MeSH Terms: conditions — Wounds and Injuries; Respiratory Insufficiency; Pneumonia, Ventilator-Associated | interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chlorhexidine gluconate: Intubated subjects transported by one air service will be treated with 5 mL chlorhexidine gluconate 0.12% applied for at least 30 seconds during helicopter transport.
  Interventions: Drug: Chlorhexidine gluconate
- Normal saline (placebo): Intubated subjects assigned transported by another air service will not have any additional treatment (in addition to usual care) during helicopter transport.

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Study solution will be applied to the oropharynx and will be distributed for 15 seconds with a swab stick. No suction will be applied for at least 30 seconds.
  Other Names: Peridex; PerioGard
  Groups: Chlorhexidine gluconate

SUMMARY:
Traumatic injury in rural America is a significant cause of morbidity and mortality, and the challenges of a rural trauma system can put patients at unique risk. Prolonged transport times to a trauma center, stopping for care at referring hospitals, and longer exposure to care-associated factors distinguish rural patients from their urban counterparts. Ventilator-associated pneumonia (VAP) is a significant risk in rural patients, increasing hospital stay, healthcare costs, and even mortality in the critically injured. The investigators propose a pilot study to test the hypothesis that a single dose of oral chlorhexidine gluconate (antiseptic) for trauma patients in the prehospital environment will decrease subsequent development of early VAP. Chlorhexidine is currently a standard therapy in intensive care units to prevent airway colonization and subsequent development of VAP. Demonstrating safety and effectiveness of prehospital infection control practices could significantly improve outcomes of traumatic injury in rural America.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >= 18 years)
* Endotracheal intubation
* Transported by air ambulance
* Traumatic injury
* Interfacility transport (no flights from scene) en route to University of Iowa Hospitals and Clinics)

Exclusion Criteria:

* Known or suspected pregnancy
* Prisoners
* Patients diagnosed with pneumonia prior to transfer
* Known allergy to chlorhexidine gluconate
* Surgical airway (tracheostomy or cricothyroidotomy)
* Massive aspiration
* Anticipated nonsurvivable injury (survival projected < 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All intubated adult patients transported by air ambulance to the University of Iowa Hospitals and Clinics in interfacility transport after traumatic injury.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical Pulmonary Infection Score (CPIS) | 48-72 hours

SECONDARY OUTCOMES:
Pneumonia - CPIS | 5 days
  This is the diagnosis of pneumonia within the first 5 days defined by CPIS score >=6.
Pneumonia - CDC | 5 days
  This is the diagnosis of pneumonia using CDC criteria within 5 days of admission.
Pneumonia - Treated | 5 days
  This is the diagnosis of pneumonia defined as antibiotic treatment of suspected pneumonia by the treating clinician.
Pneumonia - Research | 5 days
  This is the diagnosis of pneumonia within 5 days as adjudicated by 3 clinicians blinded to treatment allocation.
28-day ventilator-free days | 28 days
28-day ICU-free days | 28 days
Hospital Mortality | 28-days
Tracheostomy Rate | 28 days
Tracheal colonization | 48-72 hours
  This analysis will be completed in two ways: the raw analysis will use a chi-squared test to test the null hypothesis that the distribution of semi-quantitative tracheal colonization is the same in the two groups. A second analysis will be performed using the ordinal shift method to compare the change (shift) in the semiquantitative score between admission and 48-72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Mohr, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States